CLINICAL TRIAL: NCT05901363
Title: ERCP Plus Laparoscopic Cholecystectomy Versus Laparoscopic Common Bile Duct Exploration and Cholecystectomy for Cholecystocholedocholithiasis - The Same Operator: A Multicenter Randomized Controlled Trial
Brief Title: ERCP Plus Laparoscopic Cholecystectomy Versus Laparoscopic Common Bile Duct Exploration and Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Omar, MD, Associate professor of surgery, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVU/MED/SUR011/4/23/4/613
Record Dates: First submitted 2023-06-03; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Common Bile Duct Calculi
Keywords: Endoscopic retrograde cholangiopancreatography; laparoscopic common bile duct exploration; Laparoscopic cholecystectomy; single operator; cholecystocholedocholithiasis
MeSH Terms: conditions — Gallstones | interventions — Cholangiopancreatography, Endoscopic Retrograde; Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic retrograde cholangiopancreatography plus laparoscopic cholecystectomy (Experimental): endoscopic retrograde cholangiopancreatography plus laparoscopic cholecystectomy
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography plus laparoscopic cholecystectomy
- laparoscopic common bile duct exploration and laparoscopic cholecystectomy (Active Comparator)
  Interventions: Procedure: aparoscopic common bile duct exploration and laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography plus laparoscopic cholecystectomy — laparoscopic removal of gallbladder and endoscopic extraction of common bile duct stones
  Other Names: ERCP plus LC
  Arms: Endoscopic retrograde cholangiopancreatography plus laparoscopic cholecystectomy
Procedure: aparoscopic common bile duct exploration and laparoscopic cholecystectomy — laparoscopic removal of gallbladder and laparoscopic extraction of common bile duct stones
  Other Names: LCBDE plus LC
  Arms: laparoscopic common bile duct exploration and laparoscopic cholecystectomy

SUMMARY:
Around 10-18% of patients undergoing cholecystectomy for gallstones have common bile duct (CBD) stones. Currently, various procedures for the treatment of cholecystocholedocholithiasis are available including open cholecystectomy plus open common bile duct exploration (OC+OCBDE), laparoscopic cholecystectomy plus laparoscopic common bile duct exploration (LC+LCBDE), may be trans-cystic or trans-choledochal, and laparoscopic cholecystectomy plus endoscopic retrograde cholangiopancreatography (LC+ERCP), which may be performed pre, at, or after LC.

DETAILED DESCRIPTION:
Around 10-18% of patients undergoing cholecystectomy for gallstones have common bile duct (CBD) stones. Currently, various procedures for the treatment of cholecystocholedocholithiasis are available including open cholecystectomy plus open common bile duct exploration (OC+OCBDE), laparoscopic cholecystectomy plus laparoscopic common bile duct exploration (LC+LCBDE), may be trans-cystic or trans-choledochal, and laparoscopic cholecystectomy plus endoscopic retrograde cholangiopancreatography (LC+ERCP), which may be performed pre, at, or after LC.

Single-session treatment of gallbladder and CBD stones is safe, efficient, shortens hospital stay, and is less expensive than staged procedures.

Although there is some evidence suggesting that LCBDE may be associated with a lower rate of retained stones compared with ERCP, previous studies comparing LCBDE with ERCP and stone extraction have collectively failed to demonstrate the superiority of one approach over the other.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with cholecystocholedocholithiasis
2. American Society of Anesthesiologists (ASA) scores of I-III
3. Age 20-70 years.

Exclusion Criteria:

1. cholangitis,
2. acute biliary pancreatitis,
3. suspected Mirizzi syndrome,
4. suspected hepatobiliary malignancy,
5. perforated gallbladder,
6. biliary peritonitis,
7. intrahepatic stones,
8. pregnancy,
9. previous cholecystectomy,
10. altered anatomy such as Billroth II reconstruction or any form of Roux-en-Y reconstruction that interfere with the endoscopic approach,
11. Contraindications to laparoscopic surgery as severe liver cirrhosis or upper abdominal surgery were excluded.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
success rate | 2 years
  successful laparoscopic cholecystectomy and successful common bile duct stone extraction

SECONDARY OUTCOMES:
operative time | from 1 to 5 hours
  the overall time of the procedure
morbidity | 3 years
  any intraoperative or postoperative adverse event
mortality | 3 years
  death of patient
Hospital stay | 30 days
  the length of hospital stay from the day of admission to the day of discharge
the number of hospital readmission | 3 years
the number of postoperative intervention | 3 years
The total cost of treatment | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Omar, Principal Investigator — General Surgery Department, Faculty of Medicine, South Valley University
Locations (1):
- Mohammed Ahmed Omar, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For 1 year
Access Criteria: After publication